CLINICAL TRIAL: NCT02769416
Title: The National Center for Testing Treatments in Chronic Spinal Cord and Traumatic Brain Injury
Acronym: NCTT
Status: Enrolling by invitation | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Georgene Hergenroeder, Study Director, PI, Associate Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-15-0705
Record Dates: First submitted 2015-11-19; First posted 2016-05-11 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury; Traumatic Brain Injury
Keywords: spinal cord injury; traumatic brain injury
MeSH Terms: conditions — Spinal Cord Injuries; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood, urine, and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Cord and Traumatic Brain Injury Subjects: Patients with a history of spinal cord and/or traumatic brain injury will provide data and samples so that they may be queried for interventional studies.
  Interventions: Other: Data and sample repository
- Family Members and Healthy Volunteers: Healthy volunteer controls or family members may be enrolled for identification of genetic mutations.
  Interventions: Other: Data and sample repository

INTERVENTIONS:
Other: Data and sample repository — Subjects with spinal cord and/or traumatic brain injury, family members and healthy volunteers will provide data and samples.

SUMMARY:
The NCTT is a prospective, multicenter, observational research network for subjects with chronic spinal cord and/or chronic traumatic brain injury.

DETAILED DESCRIPTION:
Current treatment for Spinal Cord Injury and Traumatic Brain Injury focuses on stabilizing the patient and preventing secondary injury with the aim of maximizing the best chance of recovery. Most patients will show varying amounts of recovery, but, when the injury is severe, that recovery is only partial. Enrollment in the NCTT will allow for classification and characterization of injury, function, co-morbidities, secondary issues/problems, research interests and will serve as a conduit for enrollment into interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* History of spinal cord injury and/or brain injury
* Able to provide HIPAA authorization to share prior medical records/imaging
* Age 18 and older.

Exclusion Criteria:

* Life expectancy less than 6 months, vegetative state or co-existing disease or other characteristic that precludes appropriate diagnosis of spinal cord or brain injury.
* Other condition that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability or unwillingness of subject or legal guardian/representative to give informed consent (e.g., ward of the state).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic spinal cord and traumatic brain injury patients, family members, and healthy vounteers
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
International Standard Neurological Classification of Spinal Cord Injury | greater than 6 months post-injury
  functional ability (sensory and motor) for spinal cord injury subjects
Disability Rating Scale | greater than 6 months post-injury
  functional outcome scale for brain injury subjects

CONTACTS AND LOCATIONS:
Overall Officials: Georgene Hergenroeder, PhD, Principal Investigator — UTHealth
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
IPD data will not be freely available. Participating centers will share data.